CLINICAL TRIAL: NCT00810017
Title: Phase II Clinical Study Combining Trastuzumab With Etoposide in Treatment of HER2-Positive Metastatic Breast Cancer.
Brief Title: Phase 2 Study of Trastuzumab and Etoposide for Her2 Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to difficulty in accruing patients
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT_H446Us
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: HER-2 Positive Metastatic Breast Cancer
Keywords: Her2 Positive; Breast Cancer; Metastatic
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Etoposide; etoposide phosphate; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm study (Experimental): Etoposide 100mg/m2 daily x 3 days Q3W and Trastuzumab 8mg/kg loading dose then 6mg/kg, then single agent until disease progression
  Interventions: Drug: Etoposide; Drug: Trastuzumab

INTERVENTIONS:
Drug: Etoposide — etoposide 100 mg/m2 daily for 3 days every three weeks for 6 cycles
  Other Names: Eposin; Etopophos; Vepesid; VP-16
Drug: Trastuzumab — intravenous trastuzumab 8 mg/kg loading dose and then 6 mg/kg every three weeks and then single agent trastuzumab until progression of disease
  Other Names: Herceptin

SUMMARY:
This study is for women and men who have previously treated metastatic (has spread to other parts in the body), Her2- positive breast cancer. The purpose of this study is to find out what effects (good and bad) the FDA-approved drugs etoposide and trastuzumab have on this type of breast cancer and to determine if these drugs are safe to use together. This research is being done to find more effective treatment for this type of condition.

In this study, trastuzumab and etoposide will be given by intravenous infusion (IV; through a vein) on the first 3 days of every 3-week cycle. This is repeated for 6 cycles. After 6 cycles, only trastuzumab will be given until worsening of disease. In this study, a small amount of your tissue that was collected when you had surgery will be evaluated in the lab to look at genetic differences among people and how those differences may affect a response to a specific drug or medicine. This testing will look for a gene called Top2A. Previous studies suggest that people who have both the Top2A and Her2 genes respond to certain chemotherapies (anti-cancer drugs) differently from those who only have the Her2 gene.

ELIGIBILITY:
Inclusion Criteria:

* Females or males with histologic confirmation of breast carcinoma and diagnosis of metastatic breast adenocarcinoma
* Confirmed HER2 amplification by immunohistochemical staining (IHC) 3+ or FISH amplified (either primary or metastatic).
* Have had any number of prior HER2 targeted therapy containing chemotherapies for treatment of breast cancer
* Measurable extent of disease
* Life expectancy of 3 months or greater
* Patients must have adequate heart function, determined with ECHO or MUGA (ECHO preferred).
* Patients must have adequate bone marrow and organ function
* Patient of childbearing potential must be willing to use an effective means of contraception during their participation on trial
* Greater than 3 weeks from prior radiation or chemotherapy; more than 1 week from prior hormonal therapy; and more than 6 weeks from prior treatment with nitrosoureas or mitomycin.
* No serious intercurrent medical illness.
* Controlled metastatic CNS disease ≥ 3 months
* The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol.

Exclusion Criteria:

* Pregnant or nursing women
* Patients who are poor medical risk because of other non-malignant systemic disease or active, uncontrolled infection.
* Prior craniospinal radiation, or total body irradiation (TBI).
* Patients receiving G-CSF (filgrastim or pegfilgrastim) or thrombopoietin (or other platelet growth factors) within the 3 weeks prior to enrollment (erythropoietin is allowed).
* Prior chemotherapy within the last 3 weeks (last 6 weeks for nitrosureas/mitomycin).
* Prior radiation therapy within the last 3 weeks; prior radiation therapy to indicator lesion (unless objective disease recurrence or progression within the radiation portal has been documented since completion of radiation).
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Current symptoms of angina or uncontrolled arrhythmias, uncontrolled hypertension with systolic blood pressure >=170 or diastolic blood pressure >=110.
* Psychiatric illness precluding participation in study
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs, resulting in dyspnea at rest.
* Carcinomatous meningitis or CNS mets not controlled for ≥ 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M Swain, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- Washington Cancer Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm Study
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Study was terminated due to difficulties enrolling
Arm/Group | Single Arm Study
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: To Determine ORR of Trastuzumab Combined With Etoposide in Patients With HER2 Positive Metastatic Breast Cancer, and to Assess Toxicity of the Combination of Trastuzumab With Intravenous Etoposide.
Description: To determine the overall response rate
Time Frame: The best overall response is the best response recorded from the start of first treatment until the date of first progression or date of death from any cause whichever came first, assessed up to 24 months
Population: Study was terminated and no results were collected.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 0

2. Primary Outcome: To Determine Efficacy of Trastuzumab Combined With Etoposide in Patients With HER2-positive Metastatic Breast Cancer, and to Assess Toxicity of the Combination of Trastuzumab With Intravenous Etoposide.
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Time Frame: From the start of first treatment until unacceptable toxicity or date of death, whichever came first, over 24 months
Population: Study was terminated and no results were collected.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 0

3. Secondary Outcome: Determine Duration of Response
Description: Stable disease
Time Frame: Stable disease is measured from the start of the treatment until the criteria for progression are met, assessed by CT scans at a minimum interval of 8 weeks over 5 years
Population: Study was terminated and no results were collected.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 0

4. Secondary Outcome: Determine Duration of Response
Description: Time to disease progression
Time Frame: Time to disease progression is defined as time from registration date to the date of documented disease progression or death on study, whichever occurs first for 5 years
Population: Study was terminated and no results were collected.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 0

5. Secondary Outcome: Determine Duration of Response
Description: The duration of overall response will be measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started. The duration of overall CR is measured from the time measurements are met for CR until the first date that recurrent disease is objectively documented
Time Frame: The progression-free survival rate is defined as the percentage of patients who are without disease progression while on the study treatment at the end of study, over 5 years
Population: Study was terminated and no results were collected.
Arm/Group | Single Arm Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study was terminated and no results were collected.
Description: Study was terminated and no results were collected.
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No